CLINICAL TRIAL: NCT03819569
Title: GRADE-SRM: Genomic Risk Assessment and Decisional Evaluation for Small Renal Masses
Acronym: GRADE-SRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LCCC 1834
Record Dates: First submitted 2018-11-29; First posted 2019-01-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Small Renal Mass; Kidney Tumor
Keywords: genomic risk assessment; small renal mass
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: non-randomized, comparative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biopsy (Active Comparator): Subjects receive a renal cell biopsy prior to making a decision about treatment
  Interventions: Procedure: Small Renal Mass Biopsy
- No Biopsy (Sham Comparator): Subjects do not receive a renal cell biopsy prior to making a decision about treatment
  Interventions: Other: No Small Renal Mass Biopsy

INTERVENTIONS:
Procedure: Small Renal Mass Biopsy — Subjects will receive a small renal mass biopsy prior to making a treatment decision
  Arms: Biopsy
Other: No Small Renal Mass Biopsy — Subjects will not receive a small renal mass biopsy prior to making a treatment decision
  Arms: No Biopsy

SUMMARY:
Purpose: The purpose of this study is to evaluate the role of renal mass biopsy on decision-making for patients presenting with clinical T1 kidney tumors. This study also incorporates integrated biomarker study to compare the genomic data obtained through biopsy tissue to genomic information from surgical data.

DETAILED DESCRIPTION:
Primary Objective

1. To compare the decisional conflict between patients who undergo renal mass biopsy during their evaluation for SRMs versus those who do not.
2. To validate the concordance of RNA sequencing (RNAseq) and genomic-based risk stratification molecular biomarkers between renal biopsy tissue and surgical (nephrectomy) specimen tissue.

Secondary objective

1. To characterize the impact of biopsy on patient reported anxiety and uncertainty, assessment of cancer care communication, and satisfaction with cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 95
* Have a small renal mass ≤7 cm on cross-sectional radiologic study evaluated at the University of North Carolina (UNC) Urology or the UNC Cancer Hospital.
* Has voluntarily provided signed informed consent to participate and HIPAA authorization for the release of personal health information
* Willing and able to complete patient-reported outcome questionnaires
* Willing to have extra cores taken for research during the standard-of-care biopsy procedure
* Willing to allow surgical specimens to be used for research
* Willing to undergo a blood draw to evaluate for circulating tumor DNA

Exclusion Criteria

* Has staging information indicating locally advanced or metastatic disease.
* Presence of transplant kidney
* Unwilling or unable to complete informed consent
* Previous biopsy of small renal mass.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Change in Decisional Conflict | Baseline, 1-3 months (before treatment)
  Decisional conflict scale between patients who undergo renal mass biopsy, and who do not will be compared. Decisional conflict scale is a validated, 16-item instrument that measures personal perceptions of decision-making. It yields a total score from 0 to 100 (higher scores indicate more decisional conflict) and sub-scores for perceptions of uncertainty, informed values clarity, support, and effectiveness in decision-making.
Receipt of nephrectomy | 1-3 months (index treatment), 2 years
  The proportion of patients undergoing nephrectomy (radical and partial nephrectomy) between patients who undergo renal mass biopsy versus those who do not will be compared.
Genomic mutations comparison | 2 years
  Molecular subtype (ccA vs ccB) and the presence of genomic mutations between the renal mass biopsy and the surgical nephrectomy specimen will be compared.

SECONDARY OUTCOMES:
Patient-reported anxiety | Baseline, 1-3 months (before treatment), 6, 12, 18, 24 months
  Patient-reported anxiety will be assessed using the Short Form PROMIS Anxiety scale. Short Form PROMIS Anxiety is a validated 4-item survey of generalized anxiety, consisting of 5 questions, each scored using a 5-point Likert scale. High scores reflect better results.
Patient-reported cancer worry | Baseline, 1-3 months (before treatment), 6, 12, 18, 24 months
  Patient-reported cancer worry will be assessed using the Brief Worry Scale which is a 4 questions assessment designed to measure the relationship between worry and an event or behavior. This study will use the brief worry scale to measure the relationship between worry and the diagnosis of a small renal mass.
Patient-Reported Risk Perception | Baseline, 1-3 months (before treatment)
  Patient-reported Risk Perception will be assessed using 2 two-question instrument to assign a numeric risk score for patients regarding incidental renal lesions, which may facilitate accurate risk comprehension.
Patient-reported uncertainty based on Short-Form Mishel Uncertainty of Illness Scale | baseline, 1-3 months (before treatment)
  Patient-reported uncertainty will be assessed using the Short-Form Mishel Uncertainty of Illness Scale which is a validated instrument that measures the patient's perception of the uncertainty of symptoms, diagnosis, treatment, and prognosis as well as the uncertainty subscale of the Decisional Conflict Scale. The scores are summed to yield a total score with a higher score indicating greater uncertainty.
Patient-reported regret about the decision | 6, 12, 18, 24 months
  Patient-reported regret about the decision will be assessed using the Decisional regret scale. Decisional Regret scale is a 5-item regret scale that measures distress or remorse after a healthcare decision. The short form consists of 5 questions, each scored using a 5-point Likert scale, indicating a number from 1 (Strongly Agree) to 5 (Strongly Disagree).
Patient-reported health-related quality of life | Baseline, 1-3 months (before treatment), 6, 12, 18, 24 months
  Patient-reported health-related quality of life will be assessed using The PROMIS Global Health scale is an 8-item, validated survey that represents five core PROMIS domains (physical function, pain, fatigue, emotional distress, social health). Higher score indicating better quality of life.
Patient reported assessment of communication in cancer care | Baseline, 1-3 months (before treatment)
  The validated 6-item Short-Form for Patient-Centered Communication-Cancer Scale. This is a validated, 6-item instrument that measures the patient's perspective on communication in cancer care. It incorporates questions relating to exchanging information, fostering relationships, making decisions, responding to emotions, enabling self-efficacy, and managing uncertainty. Each item is scored 1-5, and the overall score is an average of 6 questions, with 5 indicating the most satisfaction. A high score indicates better communication.
Receipt of any intervention (ablation, radiation therapy, nephrectomy) | 1-3 months (index treatment), 2 years
  The proportion of patients undergoing ablation, radiation therapy, nephrectomy between patients who undergo renal mass biopsy versus those who do not will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Hung J Tan, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials